CLINICAL TRIAL: NCT00078832
Title: International Breast Cancer Intervention Study
Brief Title: Anastrozole in Preventing Breast Cancer in Postmenopausal Women at Increased Risk of Breast Cancer
Acronym: IBIS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISRCTN31488319; EU-20227; EUDRACT-2004-003991-12
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: breast cancer, chemoprevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anastrozole (Experimental): anastrozole 1mg
  Interventions: Drug: anastrozole
- placebo (Placebo Comparator): anastrozole 1mg PLACEBO
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anastrozole — aromatase inhibitor
  Other Names: Arimidex
  Arms: anastrozole
Drug: placebo — Arimidex placebo
  Arms: placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. Anastrozole may be effective in preventing breast cancer.

PURPOSE: This randomized clinical trial is studying how well anastrozole works in preventing breast cancer in postmenopausal women who are at increased risk for the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of anastrozole in preventing breast cancer in postmenopausal women at increased risk for the disease.

Secondary

* Determine the role of this drug in preventing estrogen receptor-positive breast cancer in these participants.
* Determine the effect of this drug on breast cancer mortality in these participants.
* Determine the effect of this drug on other cancers, cardiovascular disease, fracture rates, and non-breast cancer deaths in these participants.
* Determine the tolerability and acceptability of side effects of this drug in these participants.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Participants are stratified according to participating center. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral anastrozole daily for 5 years.
* Arm II: Participants receive an oral placebo daily for 5 years. In both arms, treatment continues in the absence of the development of breast cancer (including ductal carcinoma in situ), a drop in the T-score below minus 4, or the occurrence of a new fragility fracture.

Participants are followed for at least a further 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ACCRUAL: A total of 3,864 participants were recruited for this study over 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets at least 1 of the relative risk factors based on age as follows:

  * 45 to 70 years of age:

    * First-degree relative who developed breast cancer at ≤ 50 years of age
    * First-degree relative who developed bilateral breast cancer
    * Two or more first- or second-degree relatives who developed breast cancer or ovarian cancer

      * Participants having both relatives who are second degree and on the opposite sides of the family must have at least one that was diagnosed at ≤ 50 years of age
    * Nulliparous (or first birth at ≥ 30 years of age) and a first-degree relative who developed breast cancer
    * Benign biopsy with proliferative disease and a first-degree relative who developed breast cancer
    * Mammographic opacity covering at least 50% of the breast in the absence of hormone replacement therapy within the past 3 months
  * 60 to 70 years of age:

    * First-degree relative with breast cancer at any age
    * Age at menopause ≥ 55 years
    * Nulliparous or age at first birth ≥ 30 years
  * 40 to 44 years of age:

    * Two or more first- or second-degree relatives who developed breast cancer or ovarian cancer at ≤ 50 years of age
    * First-degree relative with bilateral breast cancer who developed the first breast cancer at ≤ 50 years of age
    * Nulliparous (or first birth at ≥ 30 years of age) and a first-degree relative who developed breast cancer at ≤ 40 years of age
    * Benign biopsy with proliferative disease and a first-degree relative who developed breast cancer at ≤ 40 years of age
* All age groups (40 to 70 ears of age) with a 10-year risk > 5% who do not fit into the above categories are allowed

  * Clearly apparent family history AND/OR other risk factors indicating appropriate increased risk of breast cancer for age
* The following prior breast conditions are allowed (for all age groups):

  * Lobular carcinoma in situ
  * Atypical ductal or lobular hyperplasia in a benign lesion
  * Ductal carcinoma in-situ (DCIS), diagnosed within the past 6 months, and treated by mastectomy
* No evidence of breast cancer on mammogram within the past year
* Hormone receptor status:

  * For patients with prior DCIS, estrogen- or progesterone-receptor status must have been positive

    * Must have had greater than or equal to 5% positive cells

PATIENT CHARACTERISTICS:

Age

* 40 to 70

Sex

* Female

Menopausal status

* Postmenopausal, defined as at least 1 of the following:

  * Over 60 years of age
  * Bilateral oophorectomy
  * ≤ 60 years of age with a uterus and amenorrhea for at least 12 months
  * ≤ 60 years of age without a uterus and with follicle-stimulating hormone levels > 30 IU/L

Performance status

* Not specified

Life expectancy

* At least 10 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Psychologically and physically suitable to receive 5 years of anti-estrogen therapy
* No cancer within the past 5 years except non-melanoma skin cancer or carcinoma in situ of the cervix
* No evidence of osteoporosis or fragility fractures within the spine

  * Participants with a T-score > minus 4 and no more than 2 fragility fractures are allowed
* No concurrent severe disease that would place the participant at unusual risk or confound the results of the study
* No other medical condition that would preclude the ability to receive the study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior tamoxifen, raloxifene, or other selective estrogen receptor modulator (SERM) use for more than 6 months in duration unless an IBIS-I participant (must have been off trial therapy for at least 5 years.
* No concurrent tamoxifen, raloxifene, or other SERM
* No concurrent estrogen-based hormone replacement therapy
* No concurrent systemic estrogen replacement therapy, including vaginal estrogen preparations

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior prophylactic mastectomy
* No concurrent prophylactic mastectomy

Other

* More than 6 months since prior investigational drugs

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3864 (Actual)
Dates: Start 2003-09; Primary Completion 2013-12 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Development of histologically confirmed breast cancer, both invasive and non-invasive with median follow-up at 5 years | Dec 2013

SECONDARY OUTCOMES:
Breast cancer mortality with median follow-up at 10 years | Dec 2018

CONTACTS AND LOCATIONS:
Overall Officials: Jack Cuzick, PhD, Study Chair — Queen Mary University of London; Anthony Howell, Study Chair — University of Manchester
Locations (74):
- Newcastle Mater Hospital, Newcastle, New South Wales, Australia
- University Hospitals, Leuven, Belgium
- Corporacion Nacional del Cancer, Santiago, Chile
- Herlev University Hospital, Hørsholm, Denmark
- Pirkanmaa Cancer Society, Tampere, Finland
- GBG Forschungs GMBH, Frankfurt, Germany
- Department of Oncotherapy, University of Szeged, Szeged, Hungary
- Ireland (9):
  - Beaumont Hospital, Dublin, Beaumont
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin, Tallaght
  - Cork University Hospital, Cork
  - South Infirmary Victoria Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
  - University College Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
- Division of Chemoprevention, Milan, Italy
- Sir Paul Boffa Hospital, Harper Lane, Floriana, Malta
- Instituto Portugues De Oncologia, Gabinete De Estudos Clinicos, Lisbon, Portugal
- Switzerland (6):
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Ospedale Beata Vergine, Mendrisio
  - Tumor Zentrum ZeTup St. Gallen und Chur, Sankt Gallen
  - Regionalspital, Thun
- Ortaklar cad Pehlivan sok, Basak koviah ap., Istanbul, Turkey (Türkiye)
- United Kingdom (48):
  - Tameside General Hospital, Ashton-under-Lyne, England
  - Royal Bolton Hospital, Bolton, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - St. Luke's Hospital, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Frenchay Hospital, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - Broomfield Hospital, Chelmsford, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital, Chester, England
  - Essex County Hospital, Colchester, England
  - Royal Derby Hospital, Derby, England
  - Saint Margaret's Hospital,, Epping, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Frimley Park Hospital, Frimley, England
  - Conquest Hospital, Hastings, England
  - Castle Hill Hospital, Hull, England
  - Airedale General Hospital, Keighley, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's Hospital, London, England
  - Royal Marsden - London, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Singleton Hospital, Swansea, Wales
  - Aberdeen Royal Infirmary, Aberdeen
  - Lincoln County Hospital, Grantham
  - Calderdale Royal Hospital, Huddersfield
  - Royal Free and UCL Medical School, London
  - Paterson Institute for Cancer Research, Manchester
  - Northwick Park Hospital, Middlesex
  - School of Surgical & Reproductive Sciences, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Department of General Surgery Pennine Acute Hospitals NHS Trust, Oldham
  - Derriford Hospital, Plymouth
  - Cancer Clinical Trials Centre, Sheffield
  - Weston Park Hospital, Cancer Clinical Trials Centre, Department of Clinical Oncology, Sheffield
  - Princess Anne Hospital, Southampton
  - Mid Staffordshire NHS Foundation Trust, Stafford
  - Treliske Royal Cornwall Hospital, Truro
  - Wishaw General Hospital, Wishaw
  - Yeovil District Hospital, Yeovil

REFERENCES:
- [Background] Sestak I, Singh S, Cuzick J, Blake GM, Patel R, Gossiel F, Coleman R, Dowsett M, Forbes JF, Howell A, Eastell R. Changes in bone mineral density at 3 years in postmenopausal women receiving anastrozole and risedronate in the IBIS-II bone substudy: an international, double-blind, randomised, placebo-controlled trial. Lancet Oncol. 2014 Dec;15(13):1460-1468. doi: 10.1016/S1470-2045(14)71035-6. Epub 2014 Nov 11. PMID 25456365
- [Background] Jenkins VA, Ambroisine LM, Atkins L, Cuzick J, Howell A, Fallowfield LJ. Effects of anastrozole on cognitive performance in postmenopausal women: a randomised, double-blind chemoprevention trial (IBIS II). Lancet Oncol. 2008 Oct;9(10):953-61. doi: 10.1016/S1470-2045(08)70207-9. Epub 2008 Sep 1. PMID 18768369
- [Background] Sestak I, Smith SG, Howell A, Forbes JF, Cuzick J. Early participant-reported symptoms as predictors of adherence to anastrozole in the International Breast Cancer Intervention Studies II. Ann Oncol. 2018 Feb 1;29(2):504-509. doi: 10.1093/annonc/mdx713. PMID 29126161
- [Background] Cuzick J, Sestak I, Forbes JF, Dowsett M, Knox J, Cawthorn S, Saunders C, Roche N, Mansel RE, von Minckwitz G, Bonanni B, Palva T, Howell A; IBIS-II investigators. Anastrozole for prevention of breast cancer in high-risk postmenopausal women (IBIS-II): an international, double-blind, randomised placebo-controlled trial. Lancet. 2014 Mar 22;383(9922):1041-8. doi: 10.1016/S0140-6736(13)62292-8. Epub 2013 Dec 12. PMID 24333009
- See also: Clinical trial summary from Cancer Research UK Website — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-anastrozole-to-prevent-breast-cancer-in-postmenopausal-women
- See also: IBIS-II website — https://www.ibis-trials.org/thetrials/ibistrials/ibis-2-prevention